CLINICAL TRIAL: NCT05145361
Title: A Phase Ib Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of B001 in Subjects With Aquaporin-4 Antibody (AQP4-IgG) Positive Neuromyelitis Optic Spectrum Disorder (NMOSD)
Brief Title: Clinical Study of B001 Injection in Subjects With Neuromyelitis Optic Spectrum Disorder (NMOSD)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B001-103
Record Dates: First submitted 2021-11-21; First posted 2021-12-06 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: NMO Spectrum Disorder
MeSH Terms: conditions — Neuromyelitis Optica

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- B001 injection (Experimental): Subjects randomized to this arm will receive B001 twice, at day 1 and day 15, up to the end of the study.
  Interventions: Drug: B001 injection
- Placebo (Placebo Comparator): Subjects randomized to this arm will receive Placebo twice, at day 1 and day 15, up to the end of the study.
  Interventions: Biological: Placebo

INTERVENTIONS:
Drug: B001 injection — B001 injection 50mg/5mL Intravenous solution
  Arms: B001 injection
Biological: Placebo — Placebo 5mL Intravenous solution
  Arms: Placebo

SUMMARY:
The objectives of this phase Ib study are to evaluate the efficacy, safety, pharmacokinetics, pharmacodynamics and immunogenic profiles of B001 in subjects with aquaporin-4 antibody (AQP4-IgG) positive NMOSD.

ELIGIBILITY:
Inclusion Criteria:

1. NMOSD as defined by either of the following 2015 criteria with anti-AQP4 antibody (Ab) seropositive status at screening
2. Clinical evidence of at least 1 documented relapse in last 12 months prior to screening
3. Expanded Disability Status Scale (EDSS) score from 0 to 7.5 inclusive at screening
4. Age 18 to 70 years, inclusive at the time of informed consent

Exclusion Criteria:

1. Any previous treatment with anti-CD20, eculizumab, anti-BLyS monoclonal antibody (e.g., belimumab), any other treatment for prevention of multiple sclerosis (MS) relapse (e.g., interferon, natalizumab, glatiramer acetate, fingolimod, teriflunomide or dimethyl fumarate) within 6 months prior to baseline.
2. Received immunosuppression such as azathioprine, mycophenolate mofetil, methotrexate, cyclophosphamide, tacrolimus, mitoxantrone, cyclosporine A, etc, and rug therapy, biological agents such as satralizumab, tocilizumab, eculizumab, etc, 3 months prior to the first administration.
3. Evidence of serious uncontrolled concomitant diseases that may preclude participant participation, as described; Other nervous system disease, cardiovascular disease, hematologic/hematopoiesis disease, respiratory disease, muscular disease, endocrine disease, renal/urologic disease, digestive system disease, congenital or acquired severe immunodeficiency.
4. Known active infection within 3 months prior to baseline
5. Pregnancy or lactation.
6. History of severe allergic reaction to a biologic agent
7. Evidence of chronic active hepatitis B or C
8. Evidence of active tuberculosis
9. Following laboratory abnormalities at screening*:

   1. White blood cells (WBC) <4.0 x10^3/microliter (μL)
   2. Absolute neutrophil count (ANC)
   3. Absolute lymphocyte count <0.5 x10^3/μL
   4. Platelet count <80 x 10^9/ L
   5. Aspartate aminotransferase (AST) or alanine aminotransferase
10. History of drug or alcohol abuse within 6 months prior to baseline
11. Receipt of any live or live attenuated vaccine within 4 weeks prior to baseline
12. Uncontrolled systemic diseases, including hypertension that cannot be effectively controlled after treatment (systolic blood pressure ≥150 mmHg and/or diastolic blood pressure ≥100 mmHg), diabetes, gastrointestinal diseases, etc.; or the investigator believes that there is anything inappropriate reasons for selection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-04-07 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Up to 18 days.
  Measurement of DLT in all subjects.
Evaluate incidence of treatment-emergent adverse events [Safety and Tolerability]. | Up to 1 year

SECONDARY OUTCOMES:
Maximum serum concentration (Cmax) of B001. | Through study completion, up to 2 years
  To characterize the PK (Pharmacokinetics) of B001.
Time of maximum serum concentration (Tmax) of B001. | Through study completion, up to 2 years
  To characterize the PK (Pharmacokinetics) of B001.
Area under the serum concentration-time curve (AUC) of the Dosing Interval (0-14D) of B001. | Through study completion, up to 2 years
  To characterize the PK (Pharmacokinetics) of B001.
Area under the serum concentration-time curve (AUC) of the Dosing Interval (0-Last) of B001. | Through study completion, up to 2 years
  To characterize the PK (Pharmacokinetics) of B001.
Area under the serum concentration-time curve (AUC) of the Dosing Interval (0-infinity) of B001. | Through study completion, up to 2 years
  To characterize the PK (Pharmacokinetics) of B001.
Accumulation ratio of maximum serum concentration (Rac_Cmax) of B001. | Through study completion, up to 2 years
  To characterize the PK (Pharmacokinetics) of B001.
Accumulation ratio of area under the serum concentration-time curve (Rac_AUC) of the Dosing Interval (0-14D) of B001. | Through study completion, up to 2 years
  To characterize the PK (Pharmacokinetics) of B001.
Terminal rate constant(λz) of B001. | Through study completion, up to 2 years
  To characterize the PK (Pharmacokinetics) of B001.
Half-life (t1/2) of B001. | Through study completion, up to 2 years
  To characterize the PK (Pharmacokinetics) of B001.
Total clearance(CL) of B001. | Through study completion, up to 2 years
  To characterize the PK (Pharmacokinetics) of B001.
Volume of distribution(Vz) of B001. | Through study completion, up to 2 years
  To characterize the PK (Pharmacokinetics) of B001.
Percentage of area under the serum concentration-time curve (AUC 0-infinity) obtained by extrapolation (%AUCex) of B001. | Through study completion, up to 2 years
  To characterize the PK (Pharmacokinetics) of B001.
Percentage of subjects with ADA to B001 and neutralizing resistance (Nab) | Through study completion, up to 2 years
Time to First Protocol-Defined Relapse (TFR) in the Double-Blind Period | Through study completion, up to 2 years
Change in Expanded Disability Status Scale (EDSS) Score | Through study completion, up to 2 years
  The EDSS provides a total score on a scale that ranges from 0 to 10 in 0.5 increments that represent higher levels of disability. Increasing disability is reflected in an increasing EDSS score.
Time to EDSS Worsening | Through study completion, up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Dong Shi, MD,PhD, Principal Investigator — Tianjin Medical University General Hospital
Locations (4):
- China (4):
  - Beijing Tiantan Hospital Capital Medical University, Beijing, Beijing Municipality
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Tangdu hospital,fourth military medical university, Xi’an, Shanxi
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality